CLINICAL TRIAL: NCT04565236
Title: A Post Approval Commitment Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of KOVALTRY in Chinese Children, Adolescents /Adults With Severe Hemophilia A
Brief Title: A Post Approval Commitment Study to Gain More Information on How Safe and Effective KOVALTRY is in Chinese Children, Adolescents /Adults With Severe Hemophilia A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19855; 2021-003537-11 (EudraCT Number)
Record Dates: First submitted 2020-09-04; First posted 2020-09-25 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part A: PTPs <12 years of age (Experimental): Previously treated severe hemophilia A patients (PTPs) <12 years of age
  Interventions: Biological: Recombinant Factor VIII (Kovaltry, BAY81-8973) Treatment Group 1
- Part A: PTPs ≥12 to 65 years of age (Experimental): Previously treated severe hemophilia A patients (PTPs) ≥12 to 65 years of age
  Interventions: Biological: Recombinant Factor VIII (Kovaltry, BAY81-8973) Treatment Group 2
- Part B: PUPs/MTPs <6 years of age (Experimental): Previously untreated/minimally treated severe hemophilia A patients (PUPs/MTPs) <6 years of age
  Interventions: Biological: Recombinant Factor VIII (Kovaltry, BAY81-8973) Treatment Group 3

INTERVENTIONS:
Biological: Recombinant Factor VIII (Kovaltry, BAY81-8973) Treatment Group 1 — 25 to 50 IU of Kovaltry per kg body weight given via intravenous (IV) infusion twice weekly, three times weekly, or every other day according to individual requirements for 6 months.
  The dose decisions are at the discretion of the investigator.
  Arms: Part A: PTPs <12 years of age
Biological: Recombinant Factor VIII (Kovaltry, BAY81-8973) Treatment Group 2 — 12 year-old: 25 to 50 IU of Kovaltry per kg body weight given via intravenous (IV) infusion twice weekly, three times weekly, or every other day for 6 months.
  >12 year-old: 20 to 40 IU of Kovaltry per kg of body weight given via intravenous (IV) infusion two or three times per week for 6 months.
  The dose decisions are at the discretion of the investigator.
  Arms: Part A: PTPs ≥12 to 65 years of age
Biological: Recombinant Factor VIII (Kovaltry, BAY81-8973) Treatment Group 3 — 15 to 50 IU of Kovaltry per kg body weight (minimum dose: 250 IU) given via intravenous (IV) infusions at least once a week.
  The dose decisions are at the discretion of the investigator.
  Arms: Part B: PUPs/MTPs <6 years of age

SUMMARY:
The goal of this study is to gather more information on safety and efficacy of Kovaltry for the prevention and treatment of bleeds in Chinese children, adolescents/adults with severe hemophilia A. In addition, pharmacokinetic parameters of Kovaltry will be assessed in a subset of patients.

ELIGIBILITY:
Inclusion Criteria:

Part A (PTPs):

* Chinese participants with severe hemophilia A (defined as Factor VIII (FVIII): C < 1% with one- stage clotting assay documented at the time of screening)
* Currently receiving on-demand or any type of prophylaxis treatment regimen with any FVIII product
* For participants < 12 years of age, ≥ 50 exposure days (ED); for participants ≥ 12 to 65 years of age, ≥ 150 ED with any FVIII product
* No current evidence of inhibitor
* No history of FVIII inhibitor formation
* Signed informed consent

Part B (PUPs/MTPs):

* Participants must be <6 years of age at the time of their parent or legal representative's signature of informed consent on the participant's behalf
* Chinese participants with severe hemophilia A (defined as Factor VIII (FVIII): C < 1% with one- stage clotting assay documented at the time of screening)
* PUPs must have no previous exposure to any FVIII product. MTPs must have no more than 1 ED with any purified FVIII concentrate or 3 exposures with FFP or cryoprecipitate.
* MTPs must have no current evidence of inhibitor antibody as measured by the Nijmegen-modified Bethesda assay (<0.6 BU/mL) in 2 consecutive samples and must have absence of clinical signs or symptoms of decreased response to FVIII administration. Testing for the 2 negative samples must be performed by the central laboratory at least 1 week but not more than 2 weeks apart. Participants may not receive FVIII product within 72 hours prior to the collection of samples for inhibitor testing.
* PUPs and MTPs must observe a 6-month washout period if they have received subcutaneous factor substitution therapy (emicizumab).
* PUPs may be included if they will receive their first FVIII dose with KOVALTRY for treatment of first bleed and agree to start prophylaxis as part of their care. MTPs may be included if they agree to start prophylaxis as part of their care.

Exclusion Criteria:

Part A (PTPs):

* Any other bleeding disease that is different from hemophilia A (e.g. von Willebrand disease, hemophilia B)
* Platelet count < 100 000/mm^3
* Impaired renal function (serum creatinine > 2.0 mg/dL) or active liver disease (alanine aminotransferase/aspartate aminotransferase [ALT/AST] > 5x ULN)
* Human immunodeficiency virus (HIV) positive with an absolute CD4 lymphocyte cell count < 250 cells/μL
* Known hypersensitivity to the active substance, mouse or hamster protein
* Receiving chemotherapy, immune modulatory drugs other than anti-retroviral chemotherapy, or chronic use of oral or intravenous (IV) corticosteroids (> 14 days) within the last 3 months.
* Requiring any pre-medication to tolerate FVIII infusions (e.g. antihistamines)
* Currently participating in another investigational drug study, or having previously participated in a clinical study involving an investigational drug within 30 days of signing informed consent or participated in completed interventional clinical studies with BAY81-8973 (Kovaltry)
* Planned major surgery, defined as surgery with respiratory assistance and/or general anesthesia

Part B (PUPs/MTPs):

* Any other bleeding disease that is different from hemophilia A (e.g. von Willebrand disease, hemophilia B)
* Platelet count < 100 000/mm^3
* Impaired renal function (serum creatinine >2× upper limit of normal [ULN]) or active liver disease (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >5× ULN) based on screening laboratory assessments
* MTPs with history of FVIII inhibitor formation
* Known hypersensitivity to the active substance, mouse or hamster protein
* First treatment with KOVALTRY for high risk bleeding situations (e.g., surgery, intracranial bleed) or requiring intensive or prolonged treatment
* Receiving chemotherapy, immune modulatory drugs other than anti-retroviral chemotherapy, or chronic use of oral or intravenous (IV) corticosteroids (> 14 days) within the last 3 months.
* Requiring any pre-medication to tolerate FVIII infusions (e.g. antihistamines)
* Currently participating in another investigational drug study, or having previously participated in a clinical study involving an investigational drug within 30 days of signing informed consent or participated in completed interventional clinical studies with BAY 81-8973 (Kovaltry)
* Planned major surgery, defined as surgery with respiratory assistance and/or general anesthesia
* Unable to tolerate volume of blood draws required for study participation

Ages: 0 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Children's Hospital Zhejiang University School of Med, Hangzhou, Hangzhou Province
  - Shijiazhuang General Hospital, Shijiazhuang, Hebei
  - NJ Drum Tower Hospital, the Affil Hos of NJ Univ Med School, Nanjing, Jiangsu
  - 1st Affiliated hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Children's Hospital of Shanxi, Taiyuan, Shanxi
  - Chengdu Women & Children's Central Hospital, Chengdu, Sichuan
  - Peking Union Medical College Hospital CAMS, Beijing
  - Childrens Hospital of Shanghai, Shanghai

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Part A of study was conducted in multicenter in China between 22 SEP 2020 and 04 JAN 2022. The Part B of study was conducted in multicenter in China between 07 SEP 2021 and 15 MAR 2024.
Pre-assignment Details: A total of 44 subjects were enrolled in Part A of the study. Of these, 2 subjects did not pass screening and 42 subjects participated in Part A. A total of 3 participants were enrolled in Part B of the study, and all of them passed screening.
Groups:
- Part A: PTPs <12 Years: Previously treated severe hemophilia A patients (PTPs) aged below 12 years received KOVALTRY prophylaxis and treatment.
- Part A: PTPs ≥12 Years: Previously treated severe hemophilia A patients (PTPs) aged 12 to 65 years received KOVALTRY for prophylaxis and treatment.
- Part B: PUPs <6 Years: Previously untreated severe hemophilia A patients (PUPs) aged below 6 years of age received KOVALTRY for prophylaxis and treatment.
- Part B: MTPs <6 Years: Minimally treated severe hemophilia A patients (MTPs) aged below 6 years received KOVALTRY for prophylaxis and treatment.
Period: Overall Study
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years | Part B: PUPs <6 Years | Part B: MTPs <6 Years
Started | 30 | 12 | 2 | 1
Completed | 30 | 12 | 1 | 1
Not Completed | 0 | 0 | 1 | 0
Not completed — Patient/Guardian Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years | Part B: PUPs <6 Years | Part B: MTPs <6 Years | Total
Number analyzed (Participants) | 30 | 12 | 2 | 1 | 45
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (28 days-23 months) | 0 | 0 | 1 | 0 | 1
  Children (2-11 years) | 30 | 0 | 1 | 1 | 32
  Adolescents (12-17 years) | 0 | 5 | 0 | 0 | 5
  Adults (18-64 years) | 0 | 7 | 0 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 30 | 12 | 2 | 1 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 30 | 12 | 2 | 1 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Annualized Bleeding Rate (ABR) of All Bleeding Episodes During Prophylaxis Treatment in Part A
Description: Annualized number (mean +/- standard deviation) of all bleeding episodes that occurred during the prophylaxis treatment period is reported for previously treated patients (PTPs). All bleeding episodes: sum of spontaneous bleeds and trauma bleeds exclude bleeding due to surgery.
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: Bleed per year
Arm/Group | Part A: PTPs ≥12 Years | Part A: PTPs <12 Years
Number analyzed (Participants) | 12 | 30
Bleed per year | 1.86 (2.54) [lower limit 2.54] | 3.38 (4.17) [lower limit 4.17]

2. Primary Outcome: Annualized Bleeding Rate (ABR) of All Bleeding Episodes Within 48 Hours of Previous Prophylaxis Infusion in Part B
Description: Annualized number (mean +/- standard deviation) of all bleeding episodes that occurred within 48 hours of previous prophylaxis infusion is reported for previously untreated/minimally treated patients (PUPs/MTPs). All bleeding episodes: sum of spontaneous bleeds and trauma bleeds exclude bleeding due to surgery.
Time Frame: Up to 48 hours post-infusion during 6 months
Measure: Mean (Standard Deviation); unit: Bleed per year
Arm/Group | Part B: PUPs <6 Years | Part B: MTPs <6 Years
Number analyzed (Participants) | 2 | 1
Bleed per year | 0.00 (0.00) [lower limit 0.00] | 0.00 (0.00) [lower limit 0.00]

3. Secondary Outcome: Annualized Bleeding Rate (ABR) of All Bleeding Episodes Within 48 Hours of Previous Prophylaxis Infusion in Part A
Description: Annualized number (mean +/- standard deviation) of all bleeding episodes that occurred within 48 hours of previous prophylaxis infusion is reported for previously treated patients (PTPs). All bleeding episodes: sum of spontaneous bleeds and trauma bleeds exclude bleeding due to surgery.
Time Frame: Up to 48 hours post-infusion during 6 months
Measure: Mean (Standard Deviation); unit: Bleed per year
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years
Number analyzed (Participants) | 30 | 12
Bleed per year | 2.26 (3.10) [lower limit 3.10] | 1.36 (2.19) [lower limit 2.19]

4. Secondary Outcome: Annualized Bleeding Rate (ABR) of All Bleeding Episodes During Prophylaxis Treatment in Part B
Description: Annualized number (mean +/- standard deviation) of all bleeding episodes that occurred during the prophylaxis treatment period is reported for previously untreated/minimally treated patients (PUPs/MTPs). All bleeding episodes: sum of spontaneous bleeds and trauma bleeds exclude bleeding due to surgery.
Time Frame: Up to 51 exposure days
Measure: Mean (Standard Deviation); unit: Bleed per year
Arm/Group | Part B: PUPs <6 Years | Part B: MTPs <6 Years
Number analyzed (Participants) | 2 | 1
Bleed per year | 1.13 (1.60) [lower limit 1.60] | 2.05 (0) [lower limit 0]

5. Secondary Outcome: Number of Infusions Per Bleeding Episode
Description: The mean value of number of infusions for the treatment of one bleed to achieve hemostasis is reported.
Time Frame: Part A: up to 6 months; Part B: up to 51 exposure days
Measure: Mean (Standard Deviation); unit: Infusion
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years | Part B: PUPs <6 Years | Part B: MTPs <6 Years
Number analyzed (Participants) | 17 | 5 | 1 | 1
Infusion | 1.78 (2.28) [lower limit 2.28] | 1.45 (1.29) [lower limit 1.29] | 14.00 (0.00) [lower limit 0.00] | 1.00 (0.00) [lower limit 0.00]

6. Secondary Outcome: Number of Surgeries Per Physician's Assessment of Adequacy of Hemostasis in Minor Surgery
Description: For participants who underwent minor surgeries during the study, investigators were ask to assess the adequacy of hemostasis during the surgeries as excellent, good, moderate or poor. Number of surgeries per assessment is reported.
Time Frame: Part A: up to 6 months; Part B: up to 51 exposure days
Population: Participants with surgery
Measure: Number; unit: surgery
Units Other Than Participants: surgeries
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years | Part B: PUPs <6 Years | Part B: MTPs <6 Years
Number analyzed (Participants) | 2 | 1 | 0 | 1
Number analyzed (surgeries) | 2 | 2 | 0 | 0
surgery
  Total minor surgeries: number analyzed (Participants) | 2 | 1 | 0 | 0
  Total minor surgeries | 2 | 2 |  |
  Surgeries with EXCELLENT adequacy of hemostasis: number analyzed (Participants) | 2 | 1 | 0 | 0
  Surgeries with EXCELLENT adequacy of hemostasis | 2 | 2 |  |

7. Secondary Outcome: FVIII In-vivo Recovery in Part B
Description: Incremental recovery of Factor VIII (FVIII) was determined by collecting blood samples pre-infusion and 15-30 minutes after the end of the infusion. Mean recovery values at different time points are reported.
Time Frame: At baseline, Visit 6 (ED 20), unscheduled visit and final visit, up to 51 exposure days
Population: The Part B PUP participant who discontinued didn't have any measurements for recovery calculation and therefore wasn't included in recovery analysis.
Measure: Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | Part B: PUPs <6 Years | Part B: MTPs <6 Years
Number analyzed (Participants) | 1 | 1
IU/dL per IU/kg
  Baseline (Unscheduled visit for PUP) | 1.90 (0.00) | 1.86 (0.00)
  Visit 6 (ED 20) | 0.91 (0.00) | 1.22 (0.00)
  Final visit: number analyzed (Participants) | 1 | 0
  Final visit | 1.55 (0.00) |

8. Secondary Outcome: Factor VIII Inhibitor Development by the Nijmegen Bethesda Assay
Description: Number of participants who developed a positive Factor VIII (FVIII) inhibitor level (≥0.6 Bethesda unit [BU/mL]) during the study is reported.
Time Frame: Part A: up to 6 months; Part B: up to 51 exposure days
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years | Part B: PUPs <6 Years | Part B: MTPs <6 Years
Number analyzed (Participants) | 30 | 12 | 2 | 1
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant, associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly/birth defect; another medical important serious event as judged by the investigator. AEs or SAEs were considered to be treatment emergent (TEAEs or TESAEs) if they started after the first KOVALTRY infusion and up to 3 days after the last dose.
Time Frame: Part A: up to 6 months; Part B: up to 51 exposure days
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years | Part B: PUPs <6 Years | Part B: MTPs <6 Years
Number analyzed (Participants) | 30 | 12 | 2 | 1
Participants
  Any TEAE | 13 | 3 | 1 | 1
  Maximum intensity for any TEAE - Mild | 10 | 3 | 1 | 1
  Maximum intensity for any TEAE - Moderate | 2 | 0 | 0 | 0
  Maximum intensity for any TEAE - Severe | 1 | 0 | 0 | 0
  Any study drug-related TEAE | 1 | 0 | 0 | 0
  Any TESAE | 2 | 0 | 0 | 0
  TEAE with outcome death | 0 | 0 | 0 | 0

10. Other Pre Specified Outcome: Number of Participants Without Bleeding Episode
Description: Number of participants who did not experience any bleed during the prophylaxis treatment period or within 48 hours of previous prophylaxis infusion is reported.
Time Frame: During prophylaxis treatment in Part A: up to 6 months; Part B: up to 51 exposure days
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years | Part B: PUPs <6 Years | Part B: MTPs <6 Years
Number analyzed (Participants) | 30 | 12 | 2 | 1
Participants
  During prophylaxis treatment | 13 | 7 | 1 | 0
  Within 48 hours | 16 | 8 | 2 | 1

11. Other Pre Specified Outcome: Number of Bleeds Per Assessment of Response to Treatment of Bleeds
Description: Participants or caregivers were asked to assess the response to treatment of bleeds as excellent, good, moderate or poor. Number of bleeds per assessment is reported.
Time Frame: Part A: up to 6 months; Part B: up to 51 exposure days
Measure: Number; unit: Bleeds
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years | Part B: PUPs <6 Years | Part B: MTPs <6 Years
Number analyzed (Participants) | 30 | 12 | 2 | 1
Bleeds
  Total bleeds | 51 | 11 | 1 | 1
  Bleeds without response assessment to treatment | 7 | 1 | 0 | 0
  Bleeds with EXCELLENT response to treatment | 4 | 5 | 0 | 0
  Bleeds with GOOD response to treatment | 25 | 2 | 0 | 1
  Bleeds with MODERATE response to treatment | 14 | 3 | 1 | 0
  Bleeds with POOR response to treatment | 1 | 0 | 0 | 0

12. Secondary Outcome: FVIII In-vivo Recovery in Part A
Description: as for outcome 7
Time Frame: At baseline, Month 2 and final visit, up to 6 months
Measure: Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years
Number analyzed (Participants) | 30 | 12
IU/dL per IU/kg
  Baseline | 1.82 (0.26) | 2.03 (0.46)
  Month 2 | 1.86 (0.32) | 2.12 (0.42)
  Final visit | 1.85 (0.33) | 2.06 (0.37)

13. Secondary Outcome: Maximum Observed Concentration of FVIII in Plasma (Cmax) in Part A
Description: For the assessment, participants were administered a dose of 50 IU/kg KOVALTRY. Participants must have no signs or symptoms of an acute bleeding episode. For participants below 12 years, the evaluation was only performed once at baseline. For adolescents/adult participants 12 years or older, the evaluation was performed twice at baseline and at final visit.
Time Frame: at baseline for PTPs < 12 Years and at baseline and final visit (month 6) for PTPs >= 12 Years
Population: The number of analyzed participants in group "Part A: PTPs <12 years" for category "Final Visit/ Early " is 0 because no evaluation was performed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/dL
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years
Number analyzed (Participants) | 12 | 12
IU/dL
  Baseline | 95.20 (15.24) | 114.64 (15.77)
  Final Visit/ Early Termination: number analyzed (Participants) | 0 | 12
  Final Visit/ Early Termination |  | 115.95 (17.47)

14. Secondary Outcome: Area Under the Plasma Concentration of FVIII Versus Time Curve From Zero to Infinity (AUC) in Part A
Description: as for outcome 13
Time Frame: at baseline for PTPs < 12 Years and at baseline and final visit (month 6) for PTPs >= 12 Years
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*IU/dL
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years
Number analyzed (Participants) | 12 | 12
h*IU/dL
  Baseline | 1292.97 (22.87) | 1519.38 (32.38)
  Final Visit/ Early Termination: number analyzed (Participants) | 0 | 12
  Final Visit/ Early Termination |  | 1559.29 (26.16)

15. Secondary Outcome: Half-life (t1/2) of FVIII in Plasma in Part A
Description: as for outcome 13
Time Frame: at baseline for PTPs < 12 Years and at baseline and final visit (month 6) for PTPs >= 12 Years
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Part A: PTPs <12 Years | Part A: PTPs ≥12 Years
Number analyzed (Participants) | 12 | 12
Hour
  Baseline | 10.3655 (21.22) | 11.8605 (19.25)
  Final Visit/ Early Termination: number analyzed (Participants) | 0 | 12
  Final Visit/ Early Termination |  | 11.2630 (17.29)

ADVERSE EVENTS:
Time Frame: From the first infusion to three days after last infusion, an average of 6 months for Part A and 4 months for Part B. Adverse event reporting for deaths (all causes) considers all deaths that occurred at any time during the study before the last contact. Adverse event reporting for deaths (all causes) considers all deaths that occurred at any time during the study before the last contact.
Groups:
- Part A: PTPs >=12 Years: Previously treated severe hemophilia A patients (PTPs) aged 12 to 65 years received KOVALTRY for prophylaxis and treatment
Arm/Group | Part A: PTPs >=12 Years | Part A: PTPs <12 Years | Part B: PUPs <6 Years | Part B: MTPs <6 Years
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/30 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/12 | 2/30 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 3/12 | 8/30 | 1/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: PTPs >=12 Years (N=12) | Part A: PTPs <12 Years (N=30) | Part B: PUPs <6 Years (N=2) | Part B: MTPs <6 Years (N=1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: PTPs >=12 Years (N=12) | Part A: PTPs <12 Years (N=30) | Part B: PUPs <6 Years (N=2) | Part B: MTPs <6 Years (N=1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (10) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Results of ABR of treated/target joint bleeding episodes and FVIII usage are not reported as they are other pre-defined endpoints per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall ensure that any manuscripts of publications related to the study or the results of the study are provided to Bayer for review at least 60 working days before publication, during which time the PI shall maintain confidentiality. If Bayer does not make any comments within the 60 working days, the PI is free to publish. Within 60 working days, Bayer may propose amendments to the publication and reach a consensus with the PI."

DOCUMENTS (2):
  • Study Protocol (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT04565236/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT04565236/SAP_001.pdf